CLINICAL TRIAL: NCT01393080
Title: The Study of Nimotuzumab in Combination With Paclitaxel Liposome and Carboplatin (TP Regimen) for Patient With the Advanced Non-small Cell Lung Cancer( NSCLC)
Brief Title: Nimotuzumab in Combination With Paclitaxel Liposome and Carboplatin (TP Regimen) for the Advanced NSCLC Patients
Acronym: NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-IST-NSCLC-053
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2013-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: nimotuzumab; non-small cell lung cancer; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nimotuzumab; TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimotuzumab and TP regimen (Experimental): 1. TP Regimen ：Paclitaxel Liposome,135mg/m2,d1;Carbopatin（AUC=5） d2, 3 weeks/cycle, for 4 cycles.
  2. Nimotuzumab : 200mg/w, weekly, for 6 weeks; Consolidation treatment， 200mg every 2 weeks, until the end of 4 cycles of chemotherapy or the disease progression.
  Interventions: Drug: Nimotuzumab and TP regimen
- TP Regimen (Placebo Comparator): TP Regimen：Paclitaxel Liposome,135mg/m2,d1;Carbopatin（AUC=5） d2, 3 weeks/cycle, for 4 cycles.
  Interventions: Drug: TP regimen

INTERVENTIONS:
Drug: Nimotuzumab and TP regimen — 1. TP Regims：Paclitaxel Liposome,135mg/m2,d1;Carbopatin（AUC=5） d2, 3 weeks/cycle, for 4 cycles.
  2. Nimotuzumab: 200mg/w, weekly, for 6 weeks; Consolidation treatment， 200mg every 2 weeks, until the end of 4 cycles of chemotherapy or the disease progression.
  Arms: Nimotuzumab and TP regimen
Drug: TP regimen — TP Regimen：Paclitaxel Liposome,135mg/m2,d1;Carbopatin（AUC=5） d2, 3 weeks/cycle,for 4 cycles.
  Arms: TP Regimen

SUMMARY:
Nimotuzumab (hR3) is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical efficacy has been shown in adults with head and neck cancer. This study assesses the efficacy and safety of the combination of Nimotuzumab administered concomitantly with chemotherapy in patients with NSCLC. This is a randomized, muti-center sites trial of this treatment.

DETAILED DESCRIPTION:
This is a randomized, muti-center sites trial of Nimotuzumab combination with Paclitaxel Liposome and Carboplatin (TP regimen) treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the informed consent form
2. Ages from 18 to 70 years old; both male and female.
3. Pathologically and/or cytologically ① the patients of ⅢB～Ⅳstage NSCLC; ② the patients of IIIA stage NSCLC could not receive the operation or could not operate. ③ the patients of IIIA stage NSCLC are recurrent postoperation.
4. EGFR mRNA from peripheral bloods is positive by ELISA or the expression of EGFR from tumor tissue is positive by immunohistochemical staining.
5. Functions of major organs( haemogram,heart,liver,kidney)are basically normal, White blood count ≥3.5 x 109/L with neutrophils ≥1.5 x 109/L, platelet count≥100 x 109/L, and hemoglobin ≥90g/L.

   Total bilirubin ≤1.5 times upper limit of normal (ULN) range; alkaline phosphatase(ALP)≤ 2.5 times ULN, Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN, serum creatinine ≤ 1.2 times ULN .
6. With ECOG performance status 0-2;
7. Both female and male patients must use adequate methods of contraception.

Exclusion Criteria:

1. Participation other clinical trials within 1 month prior to inclusion in the trial.
2. Previous targeted treatment of TKI or EGFR antibodies prior to inclusion in the trial.
3. Previous paclitaxel liposome and carboplatin (TP) chemotherapy prior to inclusion in the trial.
4. With other serious internal diseases or uncontrolled infection;refractoriness dysentery or enterospasm, intestinal obstruction.
5. Cardiovascular diseases history (1)Uncontrollable hypertension, unstable angina, heart infarction, or congestive heart failure and arrhythmia ( happened within 12 month prior to inclusion in the trial) (2)Ischemia checked by ECG, or clinical diagnostic Heart valve disease (3)The patients of Grade II(CTC AE 3.0) of arrhythmia, myocardial ischemia, troponin T abnormality, hypertension or left ventricular ejection fraction <50%，could not include in the TP+ nimotuzumab test group;
6. With drug addition, I.e. ,drug-taking, drug-taking for long time; type B hepatitis and C hepatitis in active stage, or with AIDS.
7. Other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ, curative carcinoma of prostate.
8. With history of serious allergic or allergy.
9. Patients with less compliance
10. Pregnancy, lactation, fertility but using a prohibited contraceptive method.
11. Not fit for the clinical trial judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12months

SECONDARY OUTCOMES:
Overall survival Time | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daliang Qi, Master, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjian Medical University Cancer Institue and Hospital, Tianjin, Tianjin Municipality, China